CLINICAL TRIAL: NCT04891185
Title: Visualisation of Indocyanine Green in Primary and Interval Debulking for Ovarian Cancer
Acronym: VIPIDO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical futility
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S65525; 2021-002449-13 (EudraCT Number)
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary Debulking Surgery (Experimental)
  Interventions: Drug: Indocyanine green
- Interval Debulking Surgery (Experimental)
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Administration of the IMP: Indocyanine green, 0,25mg/kg of body weight, intravenous bolus injection

SUMMARY:
Visualise peritoneal lesions of epithelial ovarian cancer (EOC) in both primary and interval debulking surgery by using intravascular indocyanine green (ICG) and near-infrared (NIR) light. This Trial wants to investigate whether ICG can increase the visibility of peritoneal lesions and can differentiate between peritoneal implants and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. At least 18 years of age.
3. Advanced stage epithelial ovarian cancer: FIGO stage IIIb, IIIc or IV. (For FIGO staging classification, please refer to Appendix 7).
4. A biopsy or cytology confirming the presence of high-grade serous epithelial ovarian carcinoma
5. Preoperative imaging (CT and/or MRI), describing metastatic implants, as standard of care.

Exclusion Criteria:

1. Participant has a history of following diseases:

   1. Hyperthyroidism
   2. Autonomously functioning thyroid adenoma
2. Participant has an allergy or hypersensitivity for one or more of the following components:

   1. Iodine (including potassium iodine)
   2. Indocyanine green
3. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
4. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial.
5. Participation in an interventional Trial with an investigational medicinal product (IMP) or device during the surgery itself.
6. Participant has a severe renal impairment (classified as renal function<30 ml/min/1,73m2 according to CKD-EPI).
7. Participant utilises sodium bisulfite-containing heparin preparations during the day before surgery. For Belgian registered drugs, this contains:

   1. Danaparoid (Orgaran®)
   2. Other low-molecular weight heparins registered in Belgium do not contain sodium bisulfite and are not an exclusion criterion.
8. Participants requires thyroid scintigraphy utilising radioactive iodine one week after surgery.
9. A previous history of major intra-abdominal surgery with potentially major adhesions and/or distorted anatomy.
10. Participants utilises one of the interacting drugs listed in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female
Enrollment: 14 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of correct visualisation during debulking surgery with the near-infrared (NIR) fluorescence camera of peritoneal lesions of EOC in vivo by utilising ICG. | During debulking surgery

SECONDARY OUTCOMES:
Rate of diagnostic accuracy during debulking surgery with the NIR fluorescence camera of peritoneal lesions of EOC in vivo by utilising ICG. | During debulking surgery
Percentage of lesions with positive correlation between pre-operative radiographic examination(s) and the ICG signal in vivo with the NIR fluorescence camera during surgery and immediately after surgery with the pathological examination. | During debulking surgery and immediately after debulking surgery, when the pathological examination report is available.
Obtaining the tumour-to-background ratio of fluorescence in peritoneal lesions, lymph nodes and other anatomical structures during debulking surgery by utilising still images captures with the NIR fluorescence camera. | During debulking surgery
Assessment of the number and type of adverse effects, severe adverse effects and adverse reactions with the trial dose of the IMP during and immediately after the surgery. | During debulking surgery and immediately after the surgery, up to the point in time when the pathological report is available.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
According to FAIR principle will data sharing be possible after conclusion of this trial.